CLINICAL TRIAL: NCT05415059
Title: Laryngeal, Endotracheal Airway Fixator (LEAFix): In Vivo Skin Adhesion Verification Protocol
Brief Title: LEAFix Adhesion in Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SP0935
Record Dates: First submitted 2022-06-01; First posted 2022-06-10 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-03

CONDITIONS: Adhesion
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main Cohort (Other): Cohort of healthy volunteers to have device affixed
  Interventions: Device: Covatech Stoma bag material

INTERVENTIONS:
Device: Covatech Stoma bag material — Strips of Covatech Stoma bag used to asses adhesion of 3M material to be used in LEAFix device

SUMMARY:
This study compares the adhesiveness of the 3M material to be used in the final design.

DETAILED DESCRIPTION:
The material is taken from a CE marked stoma bag. Strips will be placed on to healthy volunteers on the arm and face for 10 minutes and 24 hours. A force gauge will measure the peel force. This will be compared to previous testing on metal.

Participants will also be assessed and followed up for any adverse skin issues.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Not been in a trial in last 12 weeks
* mild to no skin issues

Exclusion Criteria:

* any significant allergies
* any allergies to skin adhesive
* any medium to severe skin issues

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-08-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Adhesion after 24 hours | 24 hours
  Adhesion after 24 hours of placement inferred from peel force measured with a force gauge at 10 minutes and 24 hours measured in Newtons (N)

SECONDARY OUTCOMES:
Skin outcomes | 7 days
  Asses for any issues with adhesion to the skin with a questionnaire on day 7 - likehart scale for different skin parameters ie. degree of itchiness with 0 being none and 3 being severe

IPD SHARING:
Plan to Share IPD: No
For internal use